CLINICAL TRIAL: NCT00122655
Title: A Randomized Prospective Study Evaluating the Impact on Fat Distribution of NRTI-Sparing Regimens in Antiretroviral Experienced Patients With Lipoatrophy ANRS 108 NONUKE Study
Brief Title: Study Evaluating the Impact on Fat Distribution of Nucleoside Reverse Transcriptase Inhibitor (NRTI)-Sparing Regimens in Antiretroviral Experienced Patients With Lipoatrophy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS108 NONUKE
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections; HIV Lipodystrophy Syndrome
Keywords: HIV infections; HIV Lipodystrophy Syndrome
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome | interventions — Protease Inhibitors

INTERVENTIONS:
Drug: non-nucleoside reverse transcriptase inhibitors
Drug: nucleoside reverse transcriptase inhibitors
Drug: protease inhibitors

SUMMARY:
The aim of this trial is to evaluate the impact on fat distribution of switching to NRTI-sparing regimens in lipoatrophic antiretroviral experienced patients with complete viral suppression.

Maintenance of virological suppression and immunological factors are also assessed.

DETAILED DESCRIPTION:
Limitations on achieving complete HIV eradication render it necessary to maintain highly active antiretroviral treatment over long periods, which may lead to the development of antiretroviral-associated toxicities. The current standard-of-care HAART regimens include a backbone of 2 nucleoside reverse transcriptase inhibitors (NRTIs). Many studies have demonstrated that NRTIs particularly thymidine analogue nucleosides are important contributors to the development of lipoatrophy. This antiretroviral family inhibits also the mitochondrial gamma-DNA polymerase, which leads to mitochondrial dysfunction and side effects such as peripheral neuropathy, pancreatitis and liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females
* Confirmed laboratory diagnosis of HIV infection
* Patients receiving a 2 or 3 NRTI-containing antiretroviral treatment for at least 3 months
* Viral load below 400 copies/ml
* Patients with a clinical peripheral lipoatrophy isolated or associated with a lipohypertrophy self reported by the patient and confirmed by physical examination

Exclusion Criteria:

* Current antiretroviral therapy with 3 classes of antiretroviral therapy
* Previous virologic failure with a non-nucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI)
* Intolerance to nevirapine and efavirenz
* Acute opportunistic infection
* Diabetes
* Transaminase levels over 5 times above the upper normal limit
* Hepatitis B virus (HBV) co-infection if the patient is receiving lamivudine therapy
* Ongoing immunotherapy including interleukin-2 (IL-2) and interferon
* Pregnancy or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Evolution from inclusion to week 48 of the peripheral fat tissue measured on computed tomography (CT) scan by a volumetric fat centralized evaluation of the thighs

SECONDARY OUTCOMES:
Evolution of the viral load (VL) from inclusion to week 48 and proportion of patients with a VL over 400 copies/ml at week 48
Change in CD4 cell count between day 0 (D0) and week 48
Change in lipid profile and glucidic metabolism between D0 and week 48
Evolution of SAT/TAT and VAT/TAT between D0 and week 48

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antoine Valantin, MD, Principal Investigator — Service des Maladies Infectieuses Hopital Pitie-Salpetriere Paris; Dominique Costagliola, Study Chair — INSERM U720
Locations (1):
- Service des Maladies infectieuses et Tropicales Hopital Pitie Salpetriere, Paris, France